CLINICAL TRIAL: NCT01230762
Title: An Open Label Study of the Long-term Safety of Dapoxetine HCl in the Treatment of Rapid Ejaculation
Brief Title: An Open-Label Study of the Long-Term Safety of Dapoxetine HCl in the Treatment of Rapid Ejaculation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Responsible Party: SR DIRECTOR CLINICAL LEADER, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR005041; C-2002-014
Record Dates: First submitted 2010-10-28; First posted 2010-10-29 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-01

CONDITIONS: Ejaculation; Erectile Dysfunction; Sexual Dysfunction
Keywords: Dapoxetine, Orgasmic disorder; Premature ejaculation; Sexual dysfunction; Sexual intercourse; Ejaculation; Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction; Sexual Dysfunction, Physiological; Sexual Dysfunctions, Psychological; Premature Ejaculation; Coitus | interventions — dapoxetine

ARMS (1):
- 001 (Experimental): dapoxetine 60 mg tablet once daily as needed (prn) (with a possible dose reduction to 30 mg once daily) for up to 9 months
  Interventions: Drug: dapoxetine

INTERVENTIONS:
Drug: dapoxetine — 60 mg tablet once daily as needed (prn) (with a possible dose reduction to 30 mg once daily) for up to 9 months

SUMMARY:
The purpose of this study is to evaluate the long-term safety of dapoxetine in men with rapid ejaculation.

DETAILED DESCRIPTION:
This is a multicenter, open-label (patients and Investigators will know the name of the drug that they are receiving) study to evaluate the long-term safety and efficacy of dapoxetine therapy in adult men with premature (rapid) ejaculation (PE) who participated in 1 of 2 previous studies of dapoxetine ( ALZA Protocol C-2002-012 or C-2002-013). The length of the study will be up to 9 months. During the study, patients will be monitored for safety by review of adverse events and findings from routine laboratory tests, vital signs measurements, electrocardiograms (ECGs), and physical examinations. Oral tablets of dapoxetine (30 mg or 60 mg) will be self-administered by patients once daily, as needed, for up to 9 months. No more than 1 dose within a 24-hour period should be taken. If the 60 mg dose of dapoxetine is not well tolerated, the dose may be decreased to 30 mg dapoxetine for the remainder of the study. Patients who do not tolerate the 30 mg dose of dapoxetine should be discontinued from the study.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment within 30 days of completion of 1 of the 2 Phase 3 controlled studies (ALZA Study C-2002-012 or Study C-2002-013)
* In the opinion of the Investigator, the patient could safely continue the use of dapoxetine treatment
* Had a systolic blood pressure of <=180 mm Hg and a diastolic blood pressure <=100 mm Hg
* Agreement by patient's sexual partner (if of childbearing potential) to ensure use of a medically acceptable method of contraception for the duration of the study Exclusion Criteria:
* Currently taking any any protocol-defined prohibited medications
* Reported a diagnosis of any sexually transmitted disease, Had a new allergy or hypersensitivity to dapoxetine or other selective serotonin reuptake inhibitors
* In the opinion of the Investigator is incapable of following the study schedule for any reason

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1774 (Actual)
Dates: Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Adverse events reported | Up to 9 months
Results from physical examinations | Months 3 and 9 or termination visit
Results from vital signs measurements | Months 1, 2 and 6
Results from clinical laboratory tests | Months 1, 3, and 9 or termination visit
Results from ECGs | At the 3 month visit and the 9 month visit/Termination Visit

SECONDARY OUTCOMES:
Results from patient reported outcomes (PRO) for perception of sexual functioning | During use of dapoxetine for up to 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA

REFERENCES:
- See also: An Open-Label Study of the Long-Term Safety of Dapoxetine HCl in the Treatment of Rapid Ejaculation. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=95&filename=CR005041_CSR.pdf